CLINICAL TRIAL: NCT06299709
Title: A Phase 1, Randomized, Open-Label, 2-part Study to Evaluate the Relative Bioavailability, Food Effect, and Dose Proportionality of a Granule Formulation of Vanzacaftor in Combination With Tezacaftor and Deutivacaftor in Healthy Adult Subjects
Brief Title: A Study To Evaluate the Relative Bioavailability, Food Effect, and Dose Proportionality of a Granule Formulation of Vanzacaftor/Tezacaftor/Deutivacaftor(VNZ/TEZ/D-IVA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX23-121-012
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — deutivacaftor, tezacaftor , vanzacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: Sequence 1 (Experimental): Participants will receive VNZ/TEZ/D-IVA reference fixed dose combination (FDC) tablet in dosing period 1, then VNZ/TEZ/D-IVA test FDC granules dose level 1 in dosing period 2, and finally VNZ/TEZ/D-IVA test FDC granules dose level 2 in dosing period 3. A washout period of 14 days will be maintained between 3 dosing periods.
  Interventions: Drug: VNZ/TEZ/D-IVA
- Part A: Sequence 2 (Experimental): Participants will receive VNZ/TEZ/D-IVA test FDC granules dose level 1 in dosing period 1, then VNZ/TEZ/D-IVA test FDC granules dose level 2 in dosing period 2, and finally VNZ/TEZ/D-IVA reference FDC tablet in dosing period 3. A washout period of 14 days will be maintained between 3 dosing periods.
  Interventions: Drug: VNZ/TEZ/D-IVA
- Part A: Sequence 3 (Experimental): Participants will receive VNZ/TEZ/D-IVA test FDC granules dose level 2 in dosing period 1, then VNZ/TEZ/D-IVA reference FDC tablet in dosing period 2, and finally VNZ/TEZ/D-IVA test FDC granules dose level 1 in dosing period 3. A washout period of 14 days will be maintained between 3 dosing periods.
  Interventions: Drug: VNZ/TEZ/D-IVA
- Part B: Sequence 1 (Experimental): Participants will receive VNZ/TEZ/D-IVA test FDC granules under fasted condition in dosing period 1, then VNZ/TEZ/D-IVA test FDC granules under fed state in dosing period 2. A washout period of 18 days will be maintained between 2 dosing periods.
  Interventions: Drug: VNZ/TEZ/D-IVA
- Part B: Sequence 2 (Experimental): Participants will receive VNZ/TEZ/D-IVA test FDC granules under fed state in dosing period 1, then VNZ/TEZ/D-IVA test FDC granules under fasted condition in dosing period 2. A washout period of 18 days will be maintained between 2 dosing periods.
  Interventions: Drug: VNZ/TEZ/D-IVA

INTERVENTIONS:
Drug: VNZ/TEZ/D-IVA — FDC tablet for oral administration.
  Other Names: VX-121/VX-661/CTP-656; VX-121/VX-661/VX-561; Vanzacaftor/tezacaftor/deutivacaftor
  Arms: Part A: Sequence 1; Part A: Sequence 2; Part A: Sequence 3
Drug: VNZ/TEZ/D-IVA — FDC granules for oral administration.
  Other Names: VX-121/VX-661/CTP-656; VX-121/VX-661/VX-561; Vanzacaftor/tezacaftor/deutivacaftor

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability, food effect, and dose proportionality of a granule formulation of VNZ/TEZ/D-IVA.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2), both inclusive
* A total body weight greater than (>)50 kg

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption
* Female participants who are pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last dose of the study drug
* Male participants with a female partner who is pregnant, nursing, or planning to become pregnant during the study or within 90 days after the last dose of the study drug

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VNZ, TEZ, and D-IVA | Pre-dose up to 288 hours Post-dose
Part B: Maximum Observed Plasma Concentration (Cmax) of VNZ, TEZ, and D-IVA | Pre-dose up to 384 hours Post-dose
Part A: Area Under the Concentration Versus Time Curve (AUC) of VNZ, TEZ, and D-IVA | Pre-dose up to 288 hours Post-dose
Part B: Area Under the Concentration Versus Time Curve (AUC) of VNZ, TEZ, and D-IVA | Pre-dose up to 384 hours Post-dose

SECONDARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 42
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 36

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing